CLINICAL TRIAL: NCT05907031
Title: Personalized Brain Functional Sector-guided Continuous Theta Burst Stimulation Therapy Targeting at the Inferior Frontal Gyrus for Aphasia After Ischemic Stroke: a RCT
Brief Title: pBFS-guided cTBS Over the Inferior Frontal Gyrus for Aphasia After Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPSA02FJ30
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Ischemic; Aphasia
MeSH Terms: conditions — Ischemic Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active cTBS group (Active Comparator): active cTBS combined with speech language therapy
  Interventions: Device: active continuous Theta Burst Stimulation
- sham cTBS group (Sham Comparator): sham cTBS combined with speech language therapy
  Interventions: Device: sham continuous Theta Burst Stimulation

INTERVENTIONS:
Device: active continuous Theta Burst Stimulation — Each patient will receive two 600-pulse cTBS stimulations per day, parted by a 15-minute rest period (a total of 1200 pulses daily), for 3-week treatment, with 5 consecutive days each week.
  Arms: active cTBS group
Device: sham continuous Theta Burst Stimulation — Each patient will receive two sham 600-pulse cTBS stimulations per day, parted by a 15-minute rest period (a total of 1200 pulses daily), for 3-week treatment, with 5 consecutive days each week.
  Arms: sham cTBS group

SUMMARY:
The objective of this trial is to evaluate the effectiveness and safeness of continuous Theta Burst Stimulation (cTBS) over the right Inferior Frontal Gyrus (IFG), guided by personalized Brain Functional Sector (pBFS) technology, on language function recovery in patients with post-ischemic stroke aphasia.

DETAILED DESCRIPTION:
Increasing evidence suggests that rTMS has been effective in treating various psychological and neurological diseases, including treating post-stroke symptoms. Using the personalized brain functional sectors (pBFS) technique, investigators could precisely identify individualized brain functional networks and the personalized language-related stimulation site based on the resting-state functional MRI data. The current study proposes to conduct a double-blinded, randomized and parallel controlled design trial, to investigate the efficacy and safety of pBFS-guided personalized rTMS intervention in post-stroke aphasic patients.

Subjects will be randomly assigned to the following two groups: active continuous TBS (cTBS) group, or a sham control group. The allocation ratio will be 1:1. The stimulation protocol consisted of a 3-week treatment, with five consecutive days each week (totally 15 day-treatment) . The stimulation procedure will be assisted with real-time neuronavigation to ensure its precision.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 35 and 75 years (including 35 and 75 years).
* Meet the diagnostic criteria of acute ischemic stroke (using the 2019 American Heart Association/American Stroke Association Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke and the 2018 Chinese Society of Neurology Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke in China). All lesions should be in the left hemisphere, and the course of disease should be more than or equal to 15 days and less than or equal to 3 months .
* Meet the diagnostic criteria for aphasia according to the Chinese version of the Western Aphasia Battery (WAB), with a WAB-aphasia quotient less than 93.8.
* First onset stroke.
* Normal functioning language abilities before the stroke, with Mandarin as their native language and an educational level higher than primary school (more than 6 years' education).
* Understand the trial and be able to provide informed consent.

Exclusion Criteria:

* Combined severe dysarthria (NIHSS item 10 score ≥ 2 points);
* Aphasia caused by bilateral hemispheric stroke, brain tumors, traumatic brain injury, Parkinson's disease, motor neuron disease, or other diseases;
* Patients with implanted electronic devices such as cardiac pacemakers, cochlear implants, or other metal foreign bodies, or those with MRI contraindications such as claustrophobia or TMS treatment contraindications;
* History of epilepsy;
* Patients with severe systemic diseases such as heart, lung, liver, kidney diseases, etc., which cannot be controlled by routine medications as confirmed by laboratory tests and examinations;
* Impaired consciousness (NIHSS item 1(a) score ≥ 1 point);
* Malignant hypertension;
* Malignant tumor;
* Patients with a life expectancy of less than 1 year due to reasons other than stroke;
* Severe hearing, visual, or cognitive impairments that prevent the patient from completing the trial;
* Patients with severe depression, anxiety, or other mental illnesses that prevent them from completing the trial;
* Patients who have received other neuroregulatory treatments such as TMS or transcranial electrical stimulation within 3 months before enrollment;
* History of alcohol abuse, drug abuse, or other substance abuse;
* Patients with other abnormal test results that make them unsuitable for participating in this trial as determined by the researchers;
* Women of childbearing age who are pregnant or planning to become pregnant;
* Patients participating in other clinical trials.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 3-week therapy
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated into an Aphasia Quotient, lower scores indicate worse outcomes.

SECONDARY OUTCOMES:
Change in the Western Aphasia Battery scores | baseline, end of the 5-day therapy, end of the follow-up of 3 weeks
  The first four subsets of the WAB (Spontaneous Speech, Auditory verbal comprehension, Repetition, Naming and word finding) will be used to evaluate the participants' language ability impairments. A Chinese adapted version of WAB will be used. The scores from all four subsets will be calculated into an Aphasia Quotient, lower scores indicate worse outcomes.
Boston Diagnostic Aphasia Examination Severity Ratings | baseline，end of the 3-week therapy，end of the follow-up of 3 weeks
  The Boston Diagnostic Aphasia Examination (BDAE) Severity Ratings is a clinical tool used to evaluate the severity and type of aphasia in individuals. The assessment includes four domains: communication abilities, language content, speech sound production and response abilities. BDAE severity ratings range from level 1 to level 5, with lower scores indicating more severe aphasia.
Chinese-version Stroke and Aphasia Quality of Life Scale 39-generic version (SAQOL-39g) | baseline，end of the 3-week therapy，end of the follow-up of 3 weeks
  The SAQOL-39g is a quality of life assessment tool that is used to evaluate the impact of stroke and aphasia on a patient's quality of life. It consists of 39 items that cover a range of domains related to the patient's quality of life, such as communication, physical functioning, mood, and social support. The items are rated on a 5-point Likert scale ranging from "not at all" to "very much", with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, PhD, Study Chair — Changping Laboratory
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China